CLINICAL TRIAL: NCT03527602
Title: Enlargement of Apical Foramen in Anterior Teeth With Apical Periodontitis and Postoperative Pain and Flare-up Rate.
Brief Title: FE in Anterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isparta Military Hospital (Other)
Responsible Party: Principal Investigator, Ibrahim Ethem YAYLALI, Head of Dentistry, Isparta Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAH-5
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Pain, Postoperative; Apical Periodontitis
Keywords: Apical patency; Endodontics
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind. (Participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Endodontic treatment will be performed in maxillary anterior teeth with necrotic pulp and periapical periodontitis. Local anaesthesia will be provided (2% Novocaine with 1:80,000 epinephrine), isolation with rubber dam and standard access cavity preparation will be done.Using 2.5 % sodium hypochlorite, canal negotiation will be done. Foraminal enlargement will be achieved with rotary files in foraminal enlargement group after determining working length. Coronal flaring with # 2 and #3 Gates-Glidden drills will be done. The canals will be obturated with gutta-percha and epoxy resin sealer. The treatments will be carried out in single-visit.
  Interventions: Procedure: Foraminal enlargement
- Control (No Intervention): In the control group, no foraminal enlargement will be performed.

INTERVENTIONS:
Procedure: Foraminal enlargement — After determining the working length, a rotary file will be inserted 1 mm beyond the WL and the apical foramen will be enlarged.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether enlarging the apical foramen causes postoperative pain in maxillary anterior teeth with apical periodontitis.

DETAILED DESCRIPTION:
Foraminal enlargement (FE) is an intentional procedure that enlarges the cement canal. However, some RCTs indicate that enlarging the FE causes postoperative pain, flare-up, and destroy the apical constriction, whilst some RCTs pointed out there is no difference in terms of pain when a FE has been performed in maxillary anterior teeth with apical periodontitis. We will assess the risk of postoperative pain as risk ratio (RR). The binary (dichotomous) data: 0-44 mm: Mild or no pain; 45-100 mm: Moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

Mature permenent maxillary anterior teeth having pulpal necrosis and apical periodontitis.

Exclusion Criteria:

Systemic disorders, diabetes, pregnancy, less than 18 years of age, immunocompromised, patients who had taken antibiotics in the past 1 month, patients who had a positive history of analgesic use within the past 3 days, previously accessed teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-05 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-05 (Estimated)

PRIMARY OUTCOMES:
100-mm Visual Analog Scale (VAS). | 5 days
  The severity of pain in 12 h, 24 h, and 2, 3, 4, and 5 days according to the VAS: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
The number of patients taking an analgesic following the endodontics treatment. | 5 days
  The patients were asked to take an analgesic in the 5 days of time frame.

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim ethem yaylali, Principal Investigator — Military Hospital, Isparta
Locations (1):
- Isparta Military Hospital, Isparta, Turkey (Türkiye)